CLINICAL TRIAL: NCT04064073
Title: A Randomized, Open Label, Single / Multiple Dose, Crossover Phase 1, Study to Evaluate Drug-Drug Interaction of DWP16001 in Combination With Metformin in Healthy Male Adults
Brief Title: Study to Evaluate Drug-Drug Interaction of DWP16001 in Combination With Metformin in Healthy Male Adults (Phase 1 Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP16001102
Record Dates: First submitted 2019-08-02; First posted 2019-08-21 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Healthy
MeSH Terms: interventions — Enavogliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: DWP16001
- 2 (Experimental)
  Interventions: Drug: Metformin IR
- 3 (Experimental)
  Interventions: Drug: DWP16001+Metformin IR

INTERVENTIONS:
Drug: DWP16001 — Tablets, Oral, once daily single dose
  Arms: 1
Drug: Metformin IR — Metformin IR 1000mg, Tablets, Oral, BID for 7 days
  Arms: 2
Drug: DWP16001+Metformin IR — Tablets, Oral, once daily single dose DWP16001 Metformin IR 1000mg
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate drug-drug interaction of DWP16001 in combination with metformin IR 1000mg in Healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adults aged 19 to 50 years at the time of screening test
* 55.0 kg ≤ Body weight ≤ 90.0 kg and 18.0 ≤ Body Mass Index (BMI) ≤ 27.0
* Written consent on voluntary decision of participation prior to the screening procedure after being fully informed of and completely understanding this study
* Eligible to participate in the study at the discretion of the investigator by physical examination, laboratory test, and history taking, etc.

Exclusion Criteria:

* Current or history of clinically significant hepatic, renal, nervous, respiratory, endocrine, hemato-oncology, cardiovascular, urogenital, psychosis disorder
* Current or history of gastrointestinal disorders or prior history of gastrointestinal surgery that may affect safety and PK/PD assessment of the study drug
* Hypersensitivity or medical history of clinically significant hypersensitivity to a drug containing an ingredient of the investigational product (DWP16001), Dapagliflozin, Metformin or similar ingredient or other drugs (e.g., aspirin, antibiotics, etc.)
* Clinical laboratory test values are outside the accepted normal range at screening
* Other exclusive inclusion criteria, as defined in the protocol

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Cmax of DWP16001 | 0-72 hours
  Peak Plasma Concetration
AUClast of DWP16001 | 0-72 hours
  Area under the plasma concentration versus time curve
Cmax,ss of Metformin | 0-144 hours
  Peak Plasma Concetration at steady-state
AUCτ,ss of Metformin | 0-144 hours
  Area under the plasma concentration versus time curve at Tau, steady-state

SECONDARY OUTCOMES:
Tmax of DWP 16001, Metformin, DWP16001 Metabolites | 0-144 hours
  Time at Cmax
AUC of DWP 16001, Metformin, DWP16001 Metabolites | 0-144 hours
  Area under the plasma concentration versus time curve
T1/2 of DWP 16001, Metformin | 0-144 hours
CL/F of DWP 16001, Metformin | 0-144 hours
  Apparent total clearance of the drug from plasma after oral administration
fe of DWP 16001, DWP16001 Metabolites | 0-72 hours
  Fraction of the drug excreted into the urine
CLR of DWP 16001 | 0-144 hours
  Renal clearance of the drug from plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea